CLINICAL TRIAL: NCT05606432
Title: Examining the Effects of Live Telehealth Exercise Training on Cardiometabolic Outcomes in Wheelchair Users
Brief Title: Cardiometabolic Health Intervention Using Movement-to-Music Exercise
Acronym: CHIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jereme Wilroy, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300009718; 5R01HD111059 (NIH)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Cardiometabolic Risk Factors in Adult Wheelchair Users
Keywords: Cardiometabolic Risk Factors; Adult Wheelchair Users

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded study that conceals the group allocation from physical outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Instructor-led, one-on-one M2M exercise group
  Interventions: Other: Instructor-led, one-on-one M2M exercise group
- Group 2 (Active Comparator): Self-guided control with pre-recorded standard exercise videos
  Interventions: Other: Self-guided control with pre-recorded standard exercise videos

INTERVENTIONS:
Other: Instructor-led, one-on-one M2M exercise group — Participants will attend 3 exercise sessions per week for 24 weeks. Each session will last 15 - 40 minutes. Increasing by 5 - 10 minutes each week. Each session will last from 25 to 50 minutes by increasing 5 to 10 minutes each week. The exercise program will focus on improving cardiorespiratory fitness using a series of movement patterns accompanied by music. The program will be tailored to individuals' abilities (e.g., use of arms only vs. truck movement together; slow vs. fast tempo music). The exercise will be prescribed at a moderate intensity level (working somewhat hard with increased heart rate and breathing rate). For the follow-up phase (weeks 25-36), participants will receive the recorded M2M exercise sessions between the M2M instructors and themselves to continue to exercise for the remaining 12 weeks.
  Arms: Group 1
Other: Self-guided control with pre-recorded standard exercise videos — Participants will exercise for 36 weeks using pre-recorded exercise videos. The videos include warm-up, flexibility, muscular strength, aerobic endurance, balance, and cool-down.
  Arms: Group 2

SUMMARY:
The study aims to test the benefits of a 24-week, cardio-emphasized Movement-to-Music exercise program for reversing cardiometabolic health risk factors compared to asynchronous, standard exercise programs among 132 adult wheelchair users. The targeted cardiometabolic health factors are waist circumference, triglycerides, "good" cholesterol, glucose, and blood pressure. Additionally, a 12-week follow-up phase (weeks 25-36) is included to see whether the gains are maintained.

DETAILED DESCRIPTION:
Baseline Assessment: Participants will be asked to complete a baseline assessment. This measures physical health (e.g., cardiometabolic health factors, fat/muscle mass) and functions (e.g., muscular strength, aerobic endurance) and a series of self-reported questionnaires that are related to participant's demographics, psychosocial health (depression, sleep, fatigue), quality of life, and physical activity behaviors (volume of activity). The onsite physical tests will take approximately 2 hours to complete. The questionnaires will be completed electronically and may take up to an hour. The assessments are listed below.

PHYSICAL TEST: The physical tests will take place (1) at the UAB Research Collaborative Center (3810 Ridgeway Dr. Birmingham, AL 35209) and (2) at Lakeshore Foundation's human performance lab (4000 Ridgeway Dr. Birmingham, AL 35209).

1. Blood draw
2. Anthropometrics (weight, height, waist circumference)
3. Body composition (amount of fat mass and fat free mass) by dual x-ray absorptiometry (DXA): DXA scans will be performed to measure any changes in fat-mass and fat-free mass. X-ray scans will be performed on 3 occasions using an iDXA whole-body scanner (GE-Lunar Radiation Corporation, Madison, WI). The radiation dose is less than 1 mrem. Scans will be analyzed using CoreScan software, and muscle mass will be estimated using published equations. Trained lab staff will be available to assist with transitioning from the wheelchair to the scan platform and back again.
4. Hand grip strength: Hand-held dynamometer will be used to measure any changes in grip strength.
5. Aerobic endurance by an arm-crank ergometer and open-circuit spirometry system: Open-circuit spirometry system will be used to measure any changes in heart rate, rate of perceived exertion (i.e., how much effort you feel you are giving), and amount of air you can breathe out while performing a 20-minute, continuous arm-crank ergometer.
6. Lung strength by spirometer: Spirometer will be used to measure how much air you exhale and how quickly you exhale. You will take a deep breath and breathe out as hard as you can for several seconds into the tube.

QUESTIONNAIRES:

1. Leisure Time Physical Activity Questionnaire for Spinal Cord Injury
2. NIH PROMIS Pain Intensity Short Form
3. NIH PROMIS Pain Interference Short Form
4. NIH PROMIS Fatigue Short Form
5. NIH PROMIS Sleep Disturbance Short Form
6. NIH PROMIS 10 Global Health Items
7. NIH PROMIS Ability to Participate in Social Roles and Activities
8. NIH PROMIS Depression Short Form
9. NIH PROMIS Anxiety Short Form
10. NIH PROMIS Physical Function Form
11. Exercise Self-efficacy Scale
12. Exercise Goal-setting and Planning Scale
13. Demographics and Health History Questionnaire
14. Rapid Eating Assessment for Participants Shortened Version

Upon completing a baseline assessment, participants will be randomly assigned to one of two groups using a computer-generated code.

Group 1: Instructor-led, one-on-one exercise group (Movement-to-Music [M2M] group) Group 2: Self-guided control with pre-recorded exercise videos

Group 1: For Instructor-led, one-on-one M2M exercise group, participants will be asked to participate in 3 exercise sessions per week for 24 weeks. Each session will last from 25 minutes up to 50 minutes. Increasing by 5 to 10 minutes each week. The exercise program will focus on improving cardiorespiratory fitness using a series of movement patterns accompanied by music. The program will be tailored to individuals' abilities (e.g., use of arms only vs. truck movement together; slow vs. fast tempo music). The exercise will be prescribed at a moderate intensity level (working somewhat hard with increased heart rate and breathing rate), which will be monitored through a wearable heart rate monitor and a custom-designed, secured online application with a personal username and password. All study equipment will be provided, including a computer tablet, tablet stand, and heart rate monitor.

Data collected by the application includes exercise minutes and heart rate. For the first 8 weeks (weeks 1-8), participants will exercise 3 sessions with M2M instructors or assistant health coaches. For the second 8 weeks (weeks 9-16), participants will exercise 2 sessions with M2M instructors or assistant health coaches and 1 session by himself/herself. The first sessions of each week you attend with M2M instructors will be video-recorded and later uploaded to a private cloud. The video-recorded sessions will be used when exercising with and without assistant health coaches. For the third 8 weeks (weeks 17-24), participants will exercise 1 session with assistant health coaches and 2 sessions by himself/herself.

Upon completing the 24-week program, you will receive the recorded exercise sessions between you and the M2M instructors to continue to exercise for the remaining 12 weeks (weeks 25-36).

Group 2: For self-guided control group, you will receive a tablet, tablet stand, and a series of pre-recorded exercise videos for 36 weeks. The videos include warm-up, flexibility, muscular strength, aerobic endurance, balance, and cool-down. Participants will receive a computer tablet and tablet stand.

12-week & 24-week Follow-up Assessments: At the end of the 12- and 24-week, participants will be asked to complete the same set of physical tests and questionnaires you completed at the beginning of the study. At the end of the 36-week, participants will also be asked to complete the same questionnaires with 2 additional surveys regarding the intervention quality, which are listed below.

QUESTIONNAIRES:

15) Physical Activity Enjoyment Scale 16) 5-star rating scale about M2M Instructors (M2M group only) or pre-recorded videos (Control group only)

At the end of the 12- and 24-week study period, participants will be contacted by phone for a brief interview. This interview is to gain information about participation in the program, such as positive and negative experiences. This call will be recorded for data analysis purposes. This interview process will be conducted for only 25% of participants (n=33) for the continuous program content and delivery process improvements.

ELIGIBILITY:
Inclusion Criteria:

1. full-time or part-time use of a wheelchair device (manual wheelchair, power wheelchair, electric scooter) self-reported as the primary means of mobility
2. ≥ 2 cardiometabolic risk factor(s),
3. no contraindication to exercise as approved by a physician's medical clearance to exercise
4. age ≥18 years
5. able to use arms to exercise
6. obtaining < 90 minutes of moderate-intensity aerobic exercise per week in the last month
7. not enrolled in a structured exercise program in the past 6 months
8. able to converse and read in English.

Exclusion Criteria:

1. medically unstable to perform home exercise as determined by their physician
2. high-level tetraplegia and unable to use arms to exercise
3. no internet access was determined via self-report and internet speed test.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic indicators - hsCRP | Baseline
  Blood test Sphygmomanometer
Cardiometabolic indicators - HbA1C | Baseline
  Blood test Sphygmomanometer
Cardiometabolic indicators - fasting insulin | Baseline
  Blood test SphygmomanometerSphygmomanometer
Cardiometabolic indicators - triglycerides | Baseline
  Blood test Sphygmomanometer
Cardiometabolic indicators - cholesterol | Baseline
  Blood test Sphygmomanometer
Cardiometabolic indicators - glucose | Baseline
  Blood test Sphygmomanometer
Cardiometabolic indicators - hsCRP | 12 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - HbA1C | 12 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - fasting insulin | 12 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - triglycerides | 12 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - cholesterol | 12 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - glucose | 12 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - hsCRP | 24 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - HbA1C | 24 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - fasting insulin | 24 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - triglycerides | 24 Weeks
  Blood test Sphygmomanometer
Cardiometabolic indicators - cholesterol | 24 Weeks
  Blood test Sphygmomanometer
Body composition - DEXA | Baseline
  Dual energy X-ray absorptiometry
Body composition - DEXA | 12 Weeks
  Dual energy X-ray absorptiometry
Body composition - DEXA | 24 Weeks
  Dual energy X-ray absorptiometry
Body composition - Waist Circumference | Baseline
  Measurement of waist size
Body composition - Waist Circumference | 12 Weeks
  Measurement of waist size
Body composition - Waist Circumference | 24 Weeks
  Measurement of waist size
Body composition - Weight | baseline
  participants weight
Body composition - Weight | 12 weeks
  participants weight
Body composition - Weight | 24 weeks
  participants weight

SECONDARY OUTCOMES:
Cardiovascular capacity - Open-circuit spirometry system (ParvoMedics TrueOne 2400) | Baseline
  Open-circuit spirometry system (ParvoMedics TrueOne 2400)
Cardiovascular capacity - Open-circuit spirometry system (ParvoMedics TrueOne 2400) | 12 Weeks
  Open-circuit spirometry system (ParvoMedics TrueOne 2400)
Cardiovascular capacity - Open-circuit spirometry system (ParvoMedics TrueOne 2400) | 24 Weeks
  Open-circuit spirometry system (ParvoMedics TrueOne 2400)
Cardiovascular capacity - Polar heart rate monitor | Baseline
  Polar heart rate monitor
Cardiovascular capacity - Polar heart rate monitor | 12 Weeks
  Polar heart rate monitor
Cardiovascular capacity - Polar heart rate monitor | 24 Weeks
  Polar heart rate monitor
Cardiovascular capacity - Borg CR10 RPE Scale | Baseline
  Borg RPE Scale
Cardiovascular capacity - Borg CR10 RPE Scale | 12 Weeks
  Borg RPE Scale
Cardiovascular capacity - Borg CR10 RPE Scale | 24 Weeks
  Borg RPE Scale
Pulmonary function | Baseline
  Spirometry (forced expiratory volume over 1 second; forced vital capacity)
Pulmonary function | 12 Weeks
  Spirometry (forced expiratory volume over 1 second; forced vital capacity)
Pulmonary function | 24 Weeks
  Spirometry (forced expiratory volume over 1 second; forced vital capacity)
Muscle strength | Baseline
  Hand-held grip strength (kg)
Muscle strength | 12 Weeks
  Hand-held grip strength (kg)
Muscle strength | 24 Weeks
  Hand-held grip strength (kg)
Physical health | Baseline
  Complete NIH PROMIS online surveys
Physical health | 12 Weeks
  Complete NIH PROMIS online surveys
Physical health | 24 Weeks
  Complete NIH PROMIS online surveys
Physical health | 36 Weeks
  Complete NIH PROMIS online surveys
Physical activity | Baseline
  Complete LTPAQ-SCI online survey
Physical activity | 12 Weeks
  Complete LTPAQ-SCI online survey
Physical activity | 24 Weeks
  Complete LTPAQ-SCI online survey
Physical activity | 36 Weeks
  Complete LTPAQ-SCI online survey

CONTACTS AND LOCATIONS:
Overall Officials: Jereme Wilroy, PhD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingahm, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Rimmer JH, Lai B, Oster R, Cowan R, Young HJ, Fisher G, Kim Y, Giannone J, Wilroy JD. Cardiometabolic Health Intervention Using Music and Exercise (CHIME) Delivered via Telehealth to Wheelchair Users: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 15;14:e57423. doi: 10.2196/57423. PMID 39814364